CLINICAL TRIAL: NCT00180232
Title: An Open Clinical Trial to Assess the Influence of Newly Prescribed Aminobiphosphonates on Arterial Stiffness (Changes of the Aortal Elasticity Due to a Newly Established Aminobiphosphinate Therapy for the Treatment of Osteoporosis)
Brief Title: An Open Clinical Trial to Assess the Influence of Newly Prescribed Aminobiphosphonates on Arterial Stiffness
Status: Withdrawn | Type: Observational
Why Stopped: Clinical partner left University,
Sponsor: Technische Universität Dresden (Other)
Other Study IDs: EK160082004
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Arteriosclerosis; Osteoporosis
MeSH Terms: conditions — Arteriosclerosis; Osteoporosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients starting an aminobisphosphonate therapy due to medical reasons Broca-index: between -20 and +25% who are willing and capable to confirm written consent to enrolment after ample information has been provided

SUMMARY:
The study tries to reveal if aminobisphosphonates influence aside the bone density also the vascular status in the typical elderly patient population

DETAILED DESCRIPTION:
The subjects - starting bisphosphonate treatment due to medical reasons - will be additionally investigated as outpatients (arterial stiffness, applanation tonometry), for each subject 3 individual dates with a duration of approx. 30 min each are scheduled, prior to therapy with bisphosphonate, after 3 and 6 month of treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients starting an aminobisphosphonate therapy due to medical reasons Broca-index: between -20 and +25% who are willing and capable to confirm written consent to enrolment after ample information has been provided

Exclusion Criteria:

* patients with major cardiovascular disease patients participating in another clinical trial 1month prior to inclusion in this study patients unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients starting an aminobisphosphonate therapy due to medical reasons Broca-index: between -20 and +25%
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-04; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Siegert, MDDPharm,Phd, Principal Investigator — Technische Universität Dresden
Locations (1):
- Medizinische Fakultät der Technischen Universität Dresden, Dresden, Germany